CLINICAL TRIAL: NCT05489614
Title: A Phase I, Open-label, Single-Dose Study to Evaluate the Pharmacokinetics, Safety, and Pharmacodynamics of Olpasiran in Subjects With Normal Renal Function and Subjects With Various Degrees of Renal Impairment
Brief Title: A Study to Evaluate the Pharmacokinetics, Safety, and Pharmacodynamics of Olpasiran in Participants With Normal Renal Function and Participants With Various Degrees of Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 20220010
Record Dates: First submitted 2022-08-03; First posted 2022-08-05 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Renal Impairment
Keywords: Olpasiran; Renal Impairment; Normal Renal Function; AMG 890
MeSH Terms: conditions — Renal Insufficiency | interventions — olpasiran

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Single Dose Olpasiran Renal Impairment (Experimental): Participants will be enrolled in 1 of 5 renal function groups based on their renal impairment status, as determined by estimated glomerular filtration rate (eGFR). All participants will receive a single dose of olpasiran on Day 1.
  Interventions: Drug: Olpasiran
- Single Dose Olpasiran Normal Renal Function (Experimental): Participants with normal renal function will be enrolled and will receive a single dose of olpasiran on Day 1.
  Interventions: Drug: Olpasiran

INTERVENTIONS:
Drug: Olpasiran — Participants will receive olpasiran by subcutaneous (SC) injection.
  Other Names: AMG 890

SUMMARY:
The primary objective of this study is to evaluate the pharmacokinetics (PK) of a single dose of olpasiran in participants with normal renal function and participants with various degrees of renal impairment.

ELIGIBILITY:
Inclusion:

* Male participants or female participants of nonchildbearing potential between 18 and 75 years of age (inclusive) at the time of Screening.
* Body mass index between 18 and 40 kg/m^2 (inclusive) at the time of Screening.
* Eligible participants classified based on established need for renal replacement therapy and eGFR at Screening. Assignment will be based on eGFR at Screening.

  1. Group 1 (Normal): eGFR ≥ 90 mL/min and no history of renal disease.
  2. Group 2 (Mild): 60 ≤ eGFR ≤ 89 mL/min.
  3. Group 3 (Moderate): 30 ≤ eGFR ≤ 59 mL/min.
  4. Group 4 (Severe): 15 ≤ eGFR ≤ 29 mL/min without dialysis.
  5. Group 5 (Kidney Failure): eGFR < 15 mL/min and dialysis patients (off-dialysis).
  6. Group 6 (Kidney Failure): eGFR < 15 mL/min and dialysis patients (on-dialysis).

Exclusion:

* Active liver disease or hepatic dysfunction, defined as aspartate aminotransferase or alanine aminotransferase > 2 times the upper limit of normal.
* Clinically significant hyperkalemia (defined by serum potassium concentration as > 5.5 mEq/L for Groups 1 to 4, > 6 mEq/L for Groups 5 and 6) at Screening or Check-in.
* History of hypersensitivity, intolerance, or allergy to any drug compound, or other substance, unless approved by the Investigator (or designee) and in consultation with the Sponsor.
* Female participants with a positive pregnancy test at Screening or Check-in.
* Participant has received a dose of an investigational drug within the past 30 days or 5 halflives, whichever is longer, prior to Check-in.

Participants in Group 1 only (participants with normal renal function) are excluded if:

• A history of renal disease or renal injury as indicated by medical history or an abnormal renal function profile at Screening or Check-in.

Participants in Groups 2 to 6 (participants with varying degrees of renal impairment) are excluded if:

• A change in disease status within 30 days of Screening, as documented by the participant's medical history, deemed clinically significant by the Investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2022-09-13 (Actual); Primary Completion 2023-10-24 (Actual); Study Completion 2023-12-19 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Serum Concentration (Cmax) of Olpasiran | Predose, 0.5, 1, 3, 6, 9, 12, 24, 36, 48, 72, 96, 144 hours (postdose), Day 15, and Day 29
Area Under the Plasma Concentration-time Curve from Time Zero to the Last Quantifiable Concentration (AUClast) of Olpasiran | Predose, 0.5, 1, 3, 6, 9, 12, 24, 36, 48, 72, 96, 144 hours (postdose), Day 15, and Day 29
Area Under the Plasma Concentration-time Curve from Time Zero to Infinity (AUCinf) of Olpasiran | Predose, 0.5, 1, 3, 6, 9, 12, 24, 36, 48, 72, 96, 144 hours (postdose), Day 15, and Day 29
Dialysis Clearance of Drug From Plasma (CLD) of Olpasiran | Pre-Dialysis, 0.5, 1, 3 hours after the start of Dialysis, and immediately following the end of Dialysis, Day 1, Day 4

SECONDARY OUTCOMES:
Area Under the Effect Time Curve (AUEC) of Plasma Lipoprotein a (Lp[a]) | Screening, Day 1, Day 2, Day 4, Day 7, Day 15, Day 29, Day 57, and Day 85
Maximum Inhibitory Effect (Imax) of Plasma Lp(a) | Screening, Day 1, Day 2, Day 4, Day 7, Day 15, Day 29, Day 57, and Day 85
Time to Reach Imax of Lp(a) | Screening, Day 1, Day 2, Day 4, Day 7, Day 15, Day 29, Day 57, and Day 85
Number of Participants Who Experience an Adverse Event (AE) | Up to Day 85
Number of Participants with Clinically Significant Changes in Clinical Laboratory Evaluations | Up to Day 85
Number of Participants with Clinically Significant Changes in 12-lead Electrocardiogram (ECG) Measurements | Up to Day 85
Number of Participants with Clinically Significant Changes in Vital Signs | Up to Day 85

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (6):
- United States (6):
  - Inland Empire Clinical Trials, LLC, Rialto, California
  - CRSCA HC LLC, dba Creekside Post Acute, Yucaipa, California
  - Clinical Pharmacology Of Miami, LLC, Miami, Florida
  - Advanced Pharma CR, LLC, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - Nucleus Network - Minneapolis, Saint Paul, Minnesota

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2 ) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com